CLINICAL TRIAL: NCT02367989
Title: A Dose-response, Double-blind, Randomized, Controlled, Cross-over Trial Examining the Effect of Barley Beta-glucan on Post-prandial Glucose Response in Healthy Adults
Brief Title: Effects of Barley on Glucose Control
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Boniface Hospital (Other)
Collaborators: Agriculture and Agri-Food Canada (Other Government)
Responsible Party: Principal Investigator, Dr. Heather Blewett, Research Scientist, St. Boniface Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 1333
Record Dates: First submitted 2015-02-04; First posted 2015-02-20 (Estimated); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Healthy
Keywords: Glucose response; Insulin response; Satiety
MeSH Terms: interventions — Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Control without fibre (Placebo Comparator): Intervention: 0g barley β-glucan no fibre.
  Dose provided in waffles given as breakfast to fasting participant at 1 of 5 visits.
  Interventions: Dietary Supplement: 0g barley β-glucan no fibre
- low barley β-glucan (Experimental): Intervention: 2g barley β-glucan
  Dose provided in waffles given as breakfast to fasting participant at 1 of 5 visits.
  Interventions: Dietary Supplement: 2g barley β-glucan
- medium barley β-glucan (Experimental): Intervention: 4g barley β-glucan
  Dose provided in waffles given as breakfast to fasting participant at 1 of 5 visits.
  Interventions: Dietary Supplement: 4g barley β-glucan
- high barley β-glucan (Experimental): Intervention: 6g barley β-glucan
  Dose provided in waffles given as breakfast to fasting participant at 1 of 5 visits.
  Interventions: Dietary Supplement: 6g barley β-glucan
- control with fibre (Placebo Comparator): Intervention: 0g barley β-glucan with fibre
  Dose provided in waffles given as breakfast to fasting participant at 1 of 5 visits.
  Interventions: Dietary Supplement: 0g barley β-glucan with fibre

INTERVENTIONS:
Dietary Supplement: 0g barley β-glucan no fibre — Food containing no barley β-glucan and no additional fibre
  Arms: Control without fibre
Dietary Supplement: 2g barley β-glucan — Food containing low amounts of barley β-glucan
  Arms: low barley β-glucan
Dietary Supplement: 4g barley β-glucan — Food containing medium amounts of barley β-glucan
  Arms: medium barley β-glucan
Dietary Supplement: 6g barley β-glucan — Food containing high amounts of barley β-glucan
  Arms: high barley β-glucan
Dietary Supplement: 0g barley β-glucan with fibre — Food containing no barley β-glucan, but matches fibre content in β-glucan treatments
  Arms: control with fibre

SUMMARY:
Lifestyle modifications that include a diet high in fibre may lower the risk of developing type 2 diabetes (CDA, 2013). In this context, the presence of soluble dietary fibre in carbohydrate rich foods has been widely recognized for its effect on post-prandial glucose response (PPGR). Among these, oat and barley derived β-glucan have received tremendous attention for their biological effects, including their ability to reduce PPGR in a wide variety of food matrices (Poppitt et al, 2007). A health claim for PPGR would increase market demand for food grade barley, and help those who want to limit the rise in blood sugar after a meal choose products to meet their goals, but there are several gaps in the literature that need to be filled before a submission to Health Canada can be successful: 1) test foods in appropriate serving sizes; 2) test both the glucose and insulin response; 3) include a reference product that matches in total fibre, macronutrient, and energy profile; 4) perform dose response. The proposed study design will address all of these gaps in the current literature and take into consideration Health Canada's guidance document for health claims related to the reduction in PPGR, which sets out the criteria by which the validity of such claims will be assessed.

Hypothesis:

Barley β-glucan will reduce the PPGR in healthy participants in a dose dependent manner.

Specific objectives:

1. To determine the minimum and most effective dose of barley β-glucan in waffles on PPGR and insulin response in a cross-over, randomized, controlled clinical trial.
2. To assess the effect of barley β-glucan in waffles on appetite-related sensations using visual analog scales.
3. To demonstrate whether the test and reference products were liked or disliked similarly by participants.
4. To assess any gastrointestinal side effects from eating the test products

DETAILED DESCRIPTION:
A double-blind, randomized, controlled, cross-over study designed to examine the PPGR to barley β-glucan will be conducted at the I.H. Asper Clinical Research Institute in Winnipeg, Manitoba. A total of 24 healthy volunteers will participate in the trial. Eligible participants who have provided consent will be asked to attend 5 clinic visits in a fasted state. At each visit hey will be given 1 set of waffles to eat that contains either 0g, 2g, 4g, or 6g of barley β-glucan, 7 finger pokes to collect capillary blood, 5 questionnaires about their appetite and a questionnaire about the acceptability of the quick bread. Each visit will last approximately 2.5h and be separated by 3-14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy male or female, between the age of 18-40 years;
2. Body mass index (BMI) 18.5-30.0 kg/m2;
3. Habitually consume breakfast, lunch and dinner in the morning, mid-day and evening, respectively;
4. Willing to provide informed consent;
5. Willing/able to comply with the requirements of the study.

Exclusion Criteria:

1. Pregnant or lactating;
2. Medical history of diabetes mellitus, fasting plasma glucose ≥7.0 mmol/L, HbA1c ≥6.0%, or use of insulin or oral medication to control blood sugar;
3. Medical history of cardiovascular disease;
4. Systolic blood pressure >140 mm Hg or diastolic blood pressure >90 mm Hg;
5. Fasting plasma total cholesterol >7.8 mmol/L;
6. Fasting plasma HDL <0.9 mmol/L;
7. Fasting plasma LDL >5.0 mmol/L;
8. Fasting plasma triglycerides >2.3 mmol/L;
9. Major surgery within the last 3 months;
10. Medical history of inflammatory disease (ie. Systemic lupus erythematosis, rheumatoid arthritis, psoriasis) or use of any corticosteroid medications within 3 months;
11. Medical history of liver disease or liver dysfunction (defined as plasma AST or ALT ≥1.5 times the upper limit of normal (ULN));
12. Medical history of kidney disease or kidney dysfunction (defined as blood urea nitrogen and creatinine ≥ 1.8 times the ULN));
13. Presence of a gastrointestinal disorder, daily use of any stomach acid-lowering medications or laxatives (including fibre supplements) within the past month or antibiotic use with the past 6 weeks;
14. Active treatment for any type of cancer within 1 year prior to study start;
15. Other medical, psychiatric, or behavioral factors that in the judgment of the principal Investigator may interfere with study participation or the ability to follow the intervention protocol;
16. Shift worker (a system of employment where an individual's normal hours of work are in part, outside the period of normal working day; 6am and 8pm);
17. Smoking, use of tobacco or a nicotine replacement product (within the last 3 months);
18. Allergies to barley or wheat flour;
19. Aversion or unwillingness to eat study foods;
20. Use of any prescription or non-prescription drug, herbal or nutritional supplement known to affect glycemia;
21. Participation in another clinical trial, current or in the past 4 weeks;
22. Unstable body weight (defined as >5% change in 3 months) or actively participating in a weight loss program.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Post-prandial glucose response | 120 minutes
  Incremental area under the curve for glucose (mmol*min/L)
Post-prandial insulin response | 120 min
  Incremental area under the curve for insulin (uIU*min/mL)

SECONDARY OUTCOMES:
hunger | 120 min
  total area under the curve (AUC) using visual analog scales
fullness | 120 min
  total area under the curve (AUC) using visual analog scales
desire to eat | 120 min
  total area under the curve (AUC) using visual analog scales
prospective consumption | 120 min
  total area under the curve (AUC) using visual analog scales

OTHER OUTCOMES:
Acceptability of waffle color | 15 min
  Ratings on a scale of 1-9
Acceptability of waffle aroma | 15 min
  Ratings on a scale of 1-9
Acceptability of waffle flavor | 15 min
  Ratings on a scale of 1-9
Acceptability of waffle texture | 15 min
  Ratings on a scale of 1-9
Acceptability of waffle frequency of consumption | 15 min
  Ratings on a scale of 1-9
Gastrointestinal side effects | 120 min
  self reporting incidence of gastrointestinal effects

CONTACTS AND LOCATIONS:
Overall Officials: Heather Blewett, PhD, Principal Investigator — Agriculture and Agri-Food Canada
Locations (1):
- I.H. Asper Clinical Research Institute, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ames NP, Rhymer CR. Issues surrounding health claims for barley. J Nutr. 2008 Jun;138(6):1237S-43S. doi: 10.1093/jn/138.6.1237S. PMID 18492863
- [Background] Aziz A, Dumais L, Barber J. Health Canada's evaluation of the use of glycemic index claims on food labels. Am J Clin Nutr. 2013 Aug;98(2):269-74. doi: 10.3945/ajcn.113.061770. Epub 2013 Jun 12. PMID 23761481
- [Background] Biorklund M, van Rees A, Mensink RP, Onning G. Changes in serum lipids and postprandial glucose and insulin concentrations after consumption of beverages with beta-glucans from oats or barley: a randomised dose-controlled trial. Eur J Clin Nutr. 2005 Nov;59(11):1272-81. doi: 10.1038/sj.ejcn.1602240. PMID 16015250
- [Background] Casiraghi MC, Garsetti M, Testolin G, Brighenti F. Post-prandial responses to cereal products enriched with barley beta-glucan. J Am Coll Nutr. 2006 Aug;25(4):313-20. doi: 10.1080/07315724.2006.10719541. PMID 16943453
- [Background] Chillo S, Ranawana DV, Pratt M, Henry CJ. Glycemic response and glycemic index of semolina spaghetti enriched with barley beta-glucan. Nutrition. 2011 Jun;27(6):653-8. doi: 10.1016/j.nut.2010.07.003. Epub 2010 Sep 24. PMID 20869206
- [Background] de Graaf C, Blom WA, Smeets PA, Stafleu A, Hendriks HF. Biomarkers of satiation and satiety. Am J Clin Nutr. 2004 Jun;79(6):946-61. doi: 10.1093/ajcn/79.6.946. PMID 15159223
- [Background] Poppitt SD, van Drunen JD, McGill AT, Mulvey TB, Leahy FE. Supplementation of a high-carbohydrate breakfast with barley beta-glucan improves postprandial glycaemic response for meals but not beverages. Asia Pac J Clin Nutr. 2007;16(1):16-24. PMID 17215176
- [Background] Thondre PS, Henry CJ. Effect of a low molecular weight, high-purity beta-glucan on in vitro digestion and glycemic response. Int J Food Sci Nutr. 2011 Nov;62(7):678-84. doi: 10.3109/09637486.2011.566849. Epub 2011 May 12. PMID 21561391
- [Background] Thondre PS, Wang K, Rosenthal AJ, Henry CJ. Glycaemic response to barley porridge varying in dietary fibre content. Br J Nutr. 2012 Mar;107(5):719-24. doi: 10.1017/S0007114511003461. Epub 2011 Jul 26. PMID 21787456
- [Background] Tosh SM. Review of human studies investigating the post-prandial blood-glucose lowering ability of oat and barley food products. Eur J Clin Nutr. 2013 Apr;67(4):310-7. doi: 10.1038/ejcn.2013.25. Epub 2013 Feb 20. PMID 23422921
- [Background] Canadian Diabetes Association. Canadian diabetes association 2008 clinical practice guidelines for the prevention and management of diabetes in Canada. Canadian Journal of Diabetes. 2008;32(1).
- [Background] Canadian Diabetes Association Clinical Practice Guidelines Expert Committee; Cheng AY. Canadian Diabetes Association 2013 clinical practice guidelines for the prevention and management of diabetes in Canada. Introduction. Can J Diabetes. 2013 Apr;37 Suppl 1:S1-3. doi: 10.1016/j.jcjd.2013.01.009. Epub 2013 Mar 26. No abstract available. PMID 24070926
- [Background] Health Canada. Summary of health Canada's assessment of a health claim about barley products and blood cholesterol lowering. [Internet].; 2012. Available from: http://www.hc-sc.gc.ca/fn-an/label-etiquet/claims-reclam/assess-evalu/barley-orge-eng.php.
- [Background] European Food Safety Authority. Guidance on the scientific requirements for health claims related to appetite ratings, weight management, and blood glucose concentrations. EFSA Journal. 2012;10(3):2604.